CLINICAL TRIAL: NCT05411536
Title: The Effects of Attentional Focus Instructions on Real-time Conscious Movement Processing While Walking in a Challenging Environment for Older Adults at Risk of Falling in Hong Kong: Implications for Rehabilitation
Brief Title: Attentional Focus Instructions and Conscious Movement Processing in Older Adults
Status: Active, not recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: 15601021
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Fall Injury; Walking, Difficulty; Gait, Unsteady
Keywords: Attentional focus instructions; Conscious movement processing; Walking; Muscle efficiency; Gait parameters
MeSH Terms: conditions — Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high reinvestor group (HRG): The participants were divided into two groups, the high reinvestor group (HRG) and the low reinvestor group (LRG), using the conventional median split of their scores on the MSRS-C (Chu & Wong, 2019; Mak et al., 2020).
  Interventions: Other: Walking trials
- low reinvestor group (LRG): The participants were divided into two groups, the high reinvestor group (HRG) and the low reinvestor group (LRG), using the conventional median split of their scores on the MSRS-C (Chu & Wong, 2019; Mak et al., 2020).
  Interventions: Other: Walking trials

INTERVENTIONS:
Other: Walking trials — All participants will complete a series of walking trials. They will first be requested to perform three practice walks followed by three walking trials on a 7.4m straight level-ground firm walkway (GW) and the other three walking trials on a 7.4m straight foam walkway (FW) in a randomised order. The dimension of the foam walkway in the FW will be 8m (length), 0.8m (width), and 0.3m (height). The starting and finishing lines of the FW will be positioned at 0.3m from each side of the FW's edges. Thus, the lengths of the FW and the GW will be identical (i.e., 7.4m). Participants will be asked to walk 7.4m and stop for each walking trial.
  After a 10-minute rest break, participants will perform nine walking trials on the GW and the other nine walking trials on the FW, including three repetitions of three different attentional focus instructions (external focus [EF], internal focus [IF], and no specific focus [NF]) in the GW and FW in a randomised order.

SUMMARY:
This study aims to provide a novel scientific contribution through addressing critical knowledge gaps, examining the effects of attentional focus instructions on real-time (state) conscious movement processing propensity, gait parameters, and muscle efficiency in older adults in Hong Kong at risk of falling while walking in a challenging environment. The study results could update our scientific understanding of the mechanisms of conscious movement processing and the interventional effects of attentional focus instructions in older adults. It could ultimately enhance the methodology used for developing the most appropriate psychomotor gait re-education intervention in rehabilitation and provide clear guidelines on the exact attentional focus training that older adults require. Further, it could mitigate the effect of conscious movement processing and risk of falling in older adults.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or above;
* able to walk independently indoor for at least 20 metres without a walking aid.

Exclusion Criteria:

* a total score of less than 24 on the MMSE-C (Chiu et al., 1994; Folstein et al., 1975);
* the presence of any untreated cerebral vascular disease, Parkinson's disease, or any other major neurological deficit;
* the presence of an unstable medical condition affecting safety while walking ;
* a history of a major fall incident within the last year;
* a static visual acuity poorer than 20/40 vision (assessed using the Tumbling E eye chart).

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults (N = 106) will be recruited from different collaborating community elderly and rehabilitation centres in Hong Kong through convenience sampling. Potential participants will be screened for eligibility by the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Real-time (state) conscious movement processing propensity | Day 0
  It will be measured by the Alpha2 EEG T3-Fz coherence.
Gait speed | Day 0
  It will be measured by the 3-D motion-capture system in the unit of meter per second (m/s).
Body sway | Day 0
  It will be measured by the 3-D motion-capture system in the unit of millimeter (mm).
Stride length | Day 0
  It will be measured by the 3-D motion-capture system in the unit of meter (m).
Stride-to-stride variability | Day 0
  It will be measured by the 3-D motion-capture system by the coefficients of variation (CV).
Muscle efficiency | Day 0
  It will be measured by the surface electromyography (EMG).

SECONDARY OUTCOMES:
Walking ability | Day 0
  It will be measured by the Timed 'Up & Go' tests.
Balance ability | Day 0
  It will be measured by the Berg Balance Scale. The minimum value of the scale is 0 and the maximum value is 56. Higher score represents better balance ability.
Fear of falling | Day 0
  It will be measured by the Chinese version of the Falls Efficacy Scale International. The minimum value of the scale is 16 and the maximum value is 64. Higher score represents higher fear of falling.
Trait conscious movement processing propensity | Day 0
  It will be measured by the Chinese version of the Movement-Specific Reinvestment Scale. The minimum value of the scale is 10 and the maximum value is 60. Higher score represents higher trait conscious movement processing propensity.

CONTACTS AND LOCATIONS:
Overall Officials: Thomson Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

REFERENCES:
- [Derived] Mak TCT, Ng SSM, Leung MCY, Wong TWL. Stress-Induced Responses in Conscious Movement Processing and Walking Behaviour in Older Adults. Stress Health. 2025 Jun;41(3):e70065. doi: 10.1002/smi.70065. PMID 40522681
- [Derived] Mak TCT, Ng SSM, Chan DCL, Wong TWL. The Influence of Attentional Focus on Gait Stability and Conscious Movement Processing During Challenging Walking Conditions in Older Adults. J Gerontol B Psychol Sci Soc Sci. 2025 May 8;80(6):gbaf059. doi: 10.1093/geronb/gbaf059. PMID 40117215